CLINICAL TRIAL: NCT04389034
Title: Retrospective Data Collection Based on Patient Records and Questionaire Based Data of Therapy Results of Allergen-specific Immunotherapy With Pollinex Quattro With Tree and/or Gras Pollen Extracts and Their Mixtures
Brief Title: Influence of Specific Immunotherapy With Pollinex Quattro (Tree-/Grass Pollen) on Allergen-specific Immunoglobulin E (IgE) Levels
Status: Completed | Type: Observational
Sponsor: Allergy Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: PQ EAST V1.0
Record Dates: First submitted 2020-04-22; First posted 2020-05-15 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Rhinitis, Allergic; Respiratory Tract Infections; Allergy; Allergic Asthma; Allergic Conjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic; Respiratory Tract Infections; Hypersensitivity; Conjunctivitis, Allergic | interventions — Pollinex Quattro

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults: Patients with IgE-induced Rhinitis, Conjunctivitis and/or asthma due to tree- and/or grass pollen induced allergy
  Interventions: Drug: Pollinex Quattro with tree- and grass pollen extracts and their mixtures

INTERVENTIONS:
Drug: Pollinex Quattro with tree- and grass pollen extracts and their mixtures — retrospective analysis of patient records of allergen-specific immunotherapy

SUMMARY:
Primary goal of this non-interventional study is to evaluate the change in level of allergen-specific IgE (EAST class) after allergen-specific immunotherapy with Pollinex Quattro with tree and/or grass pollen extracts and their mixtures under medial routine at adults with tree- and/or grass-medicated pollinosis.

DETAILED DESCRIPTION:
In this non-interventional study, the change in level of allergen-specific IgE before and after 3 or more years of allergen-specific immunotherapy with Pollinex Quattro in a patient population with tree and/or grass pollen induced pollinosis and/or asthma will be analyzed. In addition, the change in medication usage, asthma status for asthmatic patients after 3, 4 or 5 years of allergen specific immunotherapy will be evaluated. Furthermore, patients will be asked for their change in quality of life after therapy end.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Diagnosis of IgE-mediated rhinitis, conjunctivitis and bronchial asthma on grass and/or tree pollen
* completed allergen-specific immunotherapy with Pollinex Quattro with tree and/or grass pollen extracts or their mixtures according to SMPC effective during immunotherapy

Exclusion Criteria:

* Contraindication according to Summary of Product Characteristics (SMPC) effective during immunotherapy
* no additional allergen-specific immunotherapy with another product than Pollinex Quattro

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Allergic patients ≥ 18 years with IgE-mediated rhinitis, conjunctivitis and bronchial asthma on grass and/or tree pollen
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Change in allergen specific IgE after allergen-specific immunotherapy | baseline, post-treatment (after at least 3 years of allergen-specific immunotherapy)
  Efficacy

SECONDARY OUTCOMES:
Change in medication usage after allergen-specific immunotherapy | baseline, post-treatment (after at least 3 years of allergen-specific immunotherapy)
  Efficacy
Change in FEV1 (forced expiratory volume at one second; measured in %) after allergen-specific immunotherapy | baseline, post-treatment (after at least 3 years of allergen-specific immunotherapy)
  Efficacy
Change in lung function resistance (measured in Kpa/l/s) after allergen-specific immunotherapy | baseline, post-treatment (after at least 3 years of allergen-specific immunotherapy)
  Efficacy
Assessment of allergic eye symptoms (itching, tearing, redness, feeling of pressure) , on a scale 0 -10 (none - severe) after allergen-specific immunotherapy | baseline, post-treatment, at least 3 years of allergen-specific immunotherapy
  Efficacy
Assessment of allergic nasal symptoms (rhinorrhea, nasal obstruction) , on a scale 0 -10 (none - severe) after allergen-specific immunotherapy | baseline, post-treatment, at least 3 years of allergen-specific immunotherapy
  Efficacy
Assessment of allergic lung/bronchial symptoms (shortness of breath, cough), on a scale 0 -10 (none - severe) after allergen-specific immunotherapy | baseline, post-treatment, at least 3 years of allergen-specific immunotherapy
  Efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Center Dr Stollewerk/Niebecker, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided